CLINICAL TRIAL: NCT04050878
Title: Analysis of Three-dimensional Modifications Caused by Full Arch Implant Supported Dental Prosthesis With a Facial Scanner
Brief Title: Three-dimensional Assessment of Facial Alterations Induced by Dental Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Implantology Institute (Other)
Collaborators: Grupo de Investigação em Bioquímica e Biologia Oral (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: II2019-07
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Soft Tissue
Keywords: Imaging, Three-Dimensional; Technology, Dental; accuracy; extra-oral scanner

STUDY DESIGN:
Intervention Model Description: Determine the modifications caused by the use of different implant-supported dental prostheses in the soft tissues of the face, mainly upper and lower lips, by the use of a facial scanner.
Masking Description: Altough it is a single arm, the obtained STL files will be identified as A and B and the outcomes assessor will not be informed which group corresponds to the patient without or with the dental prostheses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with or without dental prostheses (Experimental): The patient will be submitted to two facial scans, one with and another without the dental prostheses and the obtained datasets will be compared to assess the differences. Marks will be made in the face to allow for measurements (digital and conventional)
  Interventions: Device: Facial scanner (Bellus3D) to assess perioral alterations

INTERVENTIONS:
Device: Facial scanner (Bellus3D) to assess perioral alterations — Use of a digital caliper for conventional measurements and a facial scanner (Bellus3D) to analyse the modifications induced by the use of implant supported dental prostheses in the lip support

SUMMARY:
Validation of the use of a facial scanner for assessment of modifications caused by the use of dental prostheses and determination of discrepancies related to conventional measurements with digital caliper.

DETAILED DESCRIPTION:
3 dimensional evaluation of lip support by the use of full arch impplant supported rehabilitations with the use of a facial scannner. Determination of discrepacies between the obtained facial scan and conventional measurements made by a digital caliper on the face.

ELIGIBILITY:
Inclusion Criteria:

* Patients rehabilitated with full implant supported upper dental prostheses.

Exclusion Criteria:

* Patients without beard, facial deformities, earrings or braces.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-21 (Actual)

PRIMARY OUTCOMES:
Soft tissue changes in µm with and without implant supported dental prostheses | Both scanning procedures will be made in the same appointment upon 3 months use of delivery of the final implant supported full dental prostheses
  Differences in the perioral soft tissues with and without dental prostheses in µm

CONTACTS AND LOCATIONS:
Overall Officials: João Carames, DDS, Phd, Study Director — Implantology Institute; Duarte Marques, DDS, PhD, Principal Investigator — Implantology Institute
Locations (1):
- Instituto de Implantologia, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided